CLINICAL TRIAL: NCT05329025
Title: A Study of the Safety and Efficacy of QL1706 in Combination With Chemotherapy in First-Line Treatment of Patients With Stage IIIB/C and Stage IV Non-Small Cell Lung Cancer
Brief Title: A Study of QL1706 Combined With Chemotherapy in Advanced Non-small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL1706-201
Record Dates: First submitted 2022-04-07; First posted 2022-04-14 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Non-small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment A (Experimental): Participants with squamous cell carcinoma will receive QL1706, paclitaxel and carboplatin by intravenous (IV) injection on Day 1 of each 21-day cycle for 4 cycles in the induction treatment. In the maintenance phase, participants will be treated with QL1706 until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: QL1706
- Treatment B (Experimental): Participants with non-squamous cell carcinoma will receive QL1706, bevacizumab, pemetrexed, and carboplatin by intravenous (IV) injection on Day 1 of each 21-day cycle for 4 cycles in the induction treatment. In the maintenance phase, participants will be treated with QL1706, bevacizumab and pemetrexed until unacceptable toxicity or loss of clinical benefit.
  Interventions: Drug: QL1706

INTERVENTIONS:
Drug: QL1706 — QL1706 will be administered by IV infusion at 5mg/kg on Day 1 of each 21-day cycle until unacceptable toxicity or loss of clinical benefit.

SUMMARY:
This study will evaluate the efficacy and safety of QL1706 when given in combination with bevacizumab, paclitaxel or pemetrexed, and carboplatin in patients with Stage IIIB/C and Stage IV Non-Small Cell Lung Cancer (NSCLC). The study will be conducted in two phases: Induction Phase and Maintenance Phase.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Stage IIIB/C or IV non-squamous NSCLC Measurable disease, as defined by RECIST v1.1 Eastern Cooperative Oncology Group Performance Status of 0 or 1 Life expectancy >=3 months Adequate hematologic and organ function

Exclusion Criteria:

* History of leptomeningeal disease Uncontrolled tumor-related pain Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently) Uncontrolled or symptomatic hypercalcemia Active or history of autoimmune disease or immune deficiency History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events Adverse events Adverse events adverse events | Informed consent until disease progression or death, which ever occurs first (up to approximately 24 months)

SECONDARY OUTCOMES:
Progression Free Survival (PFS) in the intent to treat (ITT) population, as determined by the investigator | First administration until disease progression or death, which ever occurs first (up to approximately 24 months)
Objective Response Rate (ORR) in the ITT population | First administration until disease progression or death, which ever occurs first (up to approximately 24 months)
Duration of response (DOR) in the ITT population | First administration until disease progression or death, which ever occurs first (up to approximately 24 months)
Overall Survival (OS) in the ITT population | First administration until disease progression or death, which ever occurs first (up to approximately 24 months)

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Huang Y, Yang Y, Zhao Y, Zhao H, Zhou N, Zhang Y, Chen L, Zhou T, Chen G, Wu T, Lu L, Xue S, Kang X, Zhang L, Fang W. QL1706 (anti-PD-1 IgG4/CTLA-4 antibody) plus chemotherapy with or without bevacizumab in advanced non-small cell lung cancer: a multi-cohort, phase II study. Signal Transduct Target Ther. 2024 Jan 29;9(1):23. doi: 10.1038/s41392-023-01731-x. PMID 38282003